CLINICAL TRIAL: NCT01913574
Title: Pilot Study of Acupuncture to Alleviate the Upper Abdominal Pain of Cancer Patients Treated With Neurolytic Celiac Plexus Block
Brief Title: Efficacy Study of Acupuncture to Treat the Upper Abdominal Pain of Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Jin Yong Jung, Department of anesthesiolgy, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIMI-13-01-09
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture & NCPB (Experimental): The NCPB will be administered once at the start of the trial and the acupuncture will be performed 3 times per week for 2 weeks (6 times in total).
  Interventions: Device: Acupuncture; Procedure: Neurolytic celiac plexus block (NCPB)
- NCPB (Active Comparator): The NCPB alone will be applied to the patients in this group, once at the start of the trial.
  Interventions: Procedure: Neurolytic celiac plexus block (NCPB)

INTERVENTIONS:
Device: Acupuncture — Acupuncture is applied three times a week for 20 minutes for 2 weeks (total 6 sessions). 9 Acupuncture points, CV12, CV13, P6, SP4, ST36(bilateral),LI4 (bilateral), LR3 (bilateral), ST34 (bilateral), and GB21(bilateral) are used, and CV12, CV13, ST36, and LR3 are electro-stimulated.
  Arms: Acupuncture & NCPB
Procedure: Neurolytic celiac plexus block (NCPB) — An anaesthetic test is performed injecting 2ml mepivacaine. After assessing the efficacy and safety of this test, 10 ml of absolute alcohol is injected via each needle.

SUMMARY:
This study is to investigate the effectiveness of acupuncture for alleviating the upper abdominal pain of cancer patients

DETAILED DESCRIPTION:
Neurolytic celiac plexus block (NCPB) is a commonly performed procedure in patients with intractable pain due to malignancies involving the upper and mid abdomen. Recently, acupuncture is used as one of alternative interventions to treat cancer-related pains. This pilot study aims to investigate the effectiveness of pain-relief of acupuncture via comparing acupuncture plus NCPB with NCPB alone. Total 14 cancer patients with NCPB will be randomized into two groups of acupuncture and control.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Upper abdominal pain VAS ≥ 5
* Unresectable abdominal malignancy, moderate or severe abdominal pain poorly controlled with pharmacotherapy.
* All patients had advanced cancer diagnosed by histological/cytological examination
* Follow-up possible during the clinical trial
* Written informed consent voluntarily

Exclusion Criteria:

* Patient with uncorrectable coagulopathy
* Patient with allergy to local anesthesics or alcohol..
* Previous NCPB or had implanted epidural or intrathecal analgesic therapy
* Inability to lie prone
* Disease encasing the celiac plexus on computed Tomography scan
* Patients with psychiatric diseases that could have affected the study assessments
* Significant renal or hepatic disease
* Inability to comprehend or express oneself in the Korean language
* Refusal to participate in the trial or to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale(VAS) | Change from baseline to 2 weeks
  The patients will be required to document 100mm pain VAS, where '0' represents 'no pain' and '100', 'unbearable pain'. The change of pain will be reported by comparing the mean VAS before treatment, after 1 week, after 2 week, and 1 week follow-up.

SECONDARY OUTCOMES:
Analgesic drug consumption | Change from baseline to 2 weeks
  Drug consumption per day will be documented before treatment, after 1 week, after 2 week, and 1 week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Chul Seo, KMD, Ph.D, Principal Investigator — Comprehensive and Integrative Medicine Institute; Min-Ah Gwak, KMD, Ph.D, Principal Investigator — Daegu Oriental Hospital of Daegu Haany University; Seong_Hoon Park, KMD, Principal Investigator — Comprehensive and Integrative Medicine Institute
Locations (1):
- Daegu Catholic University Medical Center, Daegu, Kyungsangbukdo, South Korea